CLINICAL TRIAL: NCT03616236
Title: Buprenorphine for Probationers and Parolees: Bridging the Gap Into Treatment
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit from study sites.
Sponsor: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRI
Record Dates: First submitted 2018-07-20; First posted 2018-08-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use
MeSH Terms: interventions — Buprenorphine, Naloxone Drug Combination; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAU (Active Comparator): Participants will receive a referral to buprenorphine treatment in the community.
  Interventions: Other: Treatment as usual
- BBT (Experimental): Participants will begin buprenorphine pharmacotherapy using the MedicaSafe buprenorphine dispensing device immediately after an on-site intake at a community supervision office and continue such treatment until they are transitioned to community buprenorphine treatment
  Interventions: Drug: Buprenorphine/Naloxone

INTERVENTIONS:
Drug: Buprenorphine/Naloxone — Participants will begin buprenorphine pharmacotherapy using the MedicaSafe buprenorphine dispensing device immediately after an on-site intake at a community supervision office and continue such treatment until they are transitioned to community buprenorphine treatment
  Other Names: BBT
  Arms: BBT
Other: Treatment as usual — Participants will receive a referral to buprenorphine treatment in the community
  Other Names: TAU
  Arms: TAU

SUMMARY:
This five-year study will evaluate the effectiveness of the administration of buprenorphine bridge treatment (BBT) to probationers and parolees compared to treatment as usual (TAU), which consists of referral to a community buprenorphine treatment program.

DETAILED DESCRIPTION:
This five-year study will evaluate the effectiveness of the administration of buprenorphine bridge treatment (BBT) to probationers and parolees compared to treatment as usual (TAU), which consists of referral to a community buprenorphine treatment program. Project implementation will occur at Guilford Avenue, the primary intake unit for Baltimore City Community Supervision (Probation and Parole). The proposed study is a parallel two-group randomized controlled trial in which 160 men and 160 women with OUD on community supervision in Baltimore will be randomly assigned within community supervision status (probation or parole) and gender to one of two treatment conditions: (1) Buprenorphine Bridge Treatment (BBT): Participants will begin buprenorphine pharmacotherapy using the MedicaSafe buprenorphine dispensing device immediately after an on-site intake at a community supervision office and continue such treatment until they are transitioned to community buprenorphine treatment; or (2) Treatment as Usual (TAU): Participants will receive a referral to buprenorphine treatment in the community. Both conditions will receive information on overdose prevention. Participants will be assessed at baseline, and 1, 2, 3, 6, and 12 months post-intake using a comprehensive assessment battery. The Primary Aim: To compare the relative effectiveness of BBT to TAU in terms of: (a) illicit opioid drug test (oral saliva) results. The Secondary Aim: To examine the extent to which BBT is superior to TAU in terms of: (b) number of days receiving opioid treatment; (c) number of days using illicit opioids; (d) quality of life (i. physical health; ii. mental health); (e) HIV risk behaviors (i. sexual behavior; ii. needle use or sharing); (f) criminal activity; (g) re-arrest; and (h) re-incarceration. The proposed study is significant because the large number of probationers/parolees with OUD have limited access to an efficacious treatment, buprenorphine pharmacotherapy. The proposed study is innovative because it would be the first trial in the US assessing the effectiveness of interim buprenorphine initiated at a community supervision office compared to referral to a community treatment program. The public health impact would be widespread, as this model of care could be scaled-up throughout many areas of the US with criminal justice populations with high rates of OUD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to the conduct of any study-related procedures
2. Male or female, 18-65 years of age, inclusive
3. Be on parole or probation for at least the next 4 months
4. Have a Baltimore City address, and (5) Primary diagnosis of (DSM-5) moderate-severe opioid use disorder (at least 4 symptoms) including current use and current physiologic dependence [Note: parolees not currently physically dependent will be allowed in the study].

Exclusion Criteria:

1. Current medical condition that may prevent the participant from safely participating in the study as determined by medical evaluation
2. Current psychosis or suicidal ideation
3. Cognitive disorders that prevent the participant from passing a study enrollment quiz
4. Any pending legal action that would interrupt study participation (eg, pending incarceration, probation/parole revocation, unadjudicated charges)
5. Exposure to any investigational drug within 8 weeks of screening
6. Current use benzodiazepines (such as Valium, Xanax and other sedatives), either prescribed or illicitly obtained
7. Currently enrolled in a methadone maintenance treatment program or taking long-acting naltrexone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
opioid use | 12 months
  illicit opioid drug test (oral saliva) results

SECONDARY OUTCOMES:
treatment adherence | 12 months
  entered community based treatment
treatment adherence | 12 months
  number of days receiving opioid treatment
opioid use days | 12 months
  number of days using illicit opioids
health-related quality of life | 12 months
  physical health using the SF-12 Health Survey
health-related quality of life | 12 months
  mental health using the SF-12 Health Survey
HIV risk behaviors | 12 months
  sexual behavior using the Risk Assessment Battery (RAB)
HIV risk behaviors | 12 months
  needle use or sharing using the Risk Assessment Battery (RB)
criminal activity | 12 months
  criminal activity days
re-arrest | 12 months
  time to re-arrest
re-incarceration | 12 months
  time to re-incarceration

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Parole & Probation, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
FRI is committed to the open and timely dissemination of research outcomes. Investigators in the proposed activity recognize that promising new methods and strategies may arise during the course of the research. Fri will abide by the principles for sharing research resources as described by NIH in "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources. Working with the research community, as well as the federal funding agency, FRI will serve the scientific community at large by sharing ideas and software to ensure that new knowledge benefits society. Our goals are to disseminate new ideas so the public can benefit from discoveries, and to generate new ideas for research and education. Any data shared will be de-identified and follow the regulations set forth in applicable Human Subjects Protection Guidelines.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At completion of the study.
Access Criteria: Contact Dr. Michael Gordon Friends Research Institute